CLINICAL TRIAL: NCT04435015
Title: The Utility of Camostat Mesylate in Patients With COVID-19 Associated Coagulopathy (CAC) and Cardiovascular Complications
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: No funding
Sponsor: Yale University (Other)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Principal Investigator, Arya Mani, Professor of Medicine and of Genetics, Yale University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2000028279
Record Dates: First submitted 2020-06-16; First posted 2020-06-17 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Coagulopathy; Cardiovascular Complication; COVID-19
MeSH Terms: conditions — Hemostatic Disorders; COVID-19 | interventions — camostat; microcrystalline cellulose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Camostat mesylate 200 mg (Experimental): Participants will be given Camostat mesylate three times daily.
  Interventions: Drug: Camostat Mesylate
- Microcrystalline Cellulose (Placebo Comparator): Participants will be given placebo three times daily.
  Interventions: Drug: Microcrystalline Cellulose, NF

INTERVENTIONS:
Drug: Camostat Mesylate — Participants will be given Camostat mesylate three times daily.
  Arms: Camostat mesylate 200 mg
Drug: Microcrystalline Cellulose, NF — Participants will be given Microcrystalline Cellulose (placebo) three times daily.
  Other Names: Placebo
  Arms: Microcrystalline Cellulose

SUMMARY:
The primary aim of this study is to determine whether Camostat mesylate reduces SARS-COV-2 associated coagulopathy. Additional aims are to determine the effect of Camostat mesylate on SARS-COV-2 associated myocardial injury, to assess duration of hypoxia or intubation, to evaluate the length of intensive care unit and hospital stay, and assess mortality rates.

DETAILED DESCRIPTION:
The trial is in-patient only. Participants are identified by the hospital physicians and house staff, and contacted by research study personnel. Potential participants fulfilling inclusion criteria and not fulfilling exclusion criteria who agree to participate and sign the informed consent undergo the enrollment process. Ono Pharmaceutical, Japan, will provide Camostat mesylate tablets. The Yale New Haven Hospital research pharmacy will receive and store the drug within 15-25C range according to protocol storage requirements.

Microcrystalline Cellulose NF (PH-102) for placebo formulation will be acquired from Fagron. Empty gelatin capsules Size 0, for over-encapsulation will be acquired from Fagron. Before Ono Pharmaceutical can send the drug, an IND will be obtained from the FDA.

Principal Investigator and the Yale New Haven Hospital research pharmacy will keep accountability records for all investigational products acquired, dispensed, used and disposed. Drugs are administered by nurses. There will be no restriction on taking other medications, activities or food intake. There are two arms to the study: (a) pharmacy-formulated placebo 3 times a day (b) 200 mg Camostat mesylate to be taken three times daily. Each arm will have 100 subjects. All patients will receive treatment until discharged. Participants will be randomized equally to Camostat mesylate or identical appearing placebo using a permuted-block design with variable block size. The actual treatment assignment will be concealed from the investigators and the participants. The randomization scheme will be generated by the statistical group.

Participants have the option of refusing study drug. If the participant decides to stop the drug or blood drawing he or she would be dropped from the trial.

ELIGIBILITY:
Inclusion Criteria:

1. . Positive COVID-19 test result.
2. Diagnosis of COVID-19 associated coagulopathy and cardiac complications based on D-Dimer, fibrinogen, TnT, CTPE, ischemic EKG changes
3. Provision of informed consent. In patients with altered mental status consents can be obtained from the power of attorney.
4. Stated willingness to comply with all study procedures and availability for the duration of the study
5. Male or female, age 18 or older
6. Diagnosed with hypoxia requiring intubation or positive air pressure.
7. Diagnose with DVT/PE by ultrasound and CTPE and/or
8. Elevated D-Dimer and/or
9. Greater than 2-fold increase in TnT
10. Ischemic EKG changes with ST depression or elevation more than 1 mm in 2 consecutive leads
11. Ability to administer oral medication.

Exclusion Criteria:

1. GFR<30 mL/min
2. Severe bleeding requiring blood transfusion of drop of 5% in HCT.
3. Pregnancy or lactation
4. Known allergic reactions to components of Camostat mesylate.
5. Subjects under age 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-11 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Percent change in plasma D-Dimer | 7 days
  The sum percent change in D-Dimer over 7 days will be compared to day 1

SECONDARY OUTCOMES:
Overall Safety and adverse event | 3 months
  The first assessment on mortality and complications will be carried out 3 months after the start of the study.
Change in plasma Fibrinogen levels | 7 days
  Percent change in fibrinogen over 7 days compared to day 1
Change in plasma troponin | 7 days
  Percent change in troponin over 7 days compared to day 1
New onset cardiomyopathy | 7 days
  New onset cardiomyopathy defined by a reduction of EF by greater than 10% or less than 45% will be measured
Duration of intubation | 7 days
  Days with hypoxia (Room Air O2 Sat<93%) or days intubated
Length of stay in the intensive care unit | 28 days
  The number of days in the intensive care unit
Time to discharge from hospital | 30 days
  The number of days since admission to discharge
Occurrence of major adverse cardiovascular events | 7 days
  The ocurrence of major adverse cardiovascular events (MACE): MI, stroke, CHF, PCI, death from cardiovascular disease will be studied.

CONTACTS AND LOCATIONS:
Overall Officials: Arya Mani, MD, Principal Investigator — Yale University

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR
Time Frame: Study protocol and clinical study report will be shared 1 year after completion of the study